CLINICAL TRIAL: NCT03690297
Title: Linked Color Imaging (LCI) Versus Standard White-light Colonoscopy for Colorectal Adenoma Detection: a Multicenter, Randomized, Trial
Brief Title: Linked Color Imaging (LCI) for Colorectal Adenoma Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Franco Radaelli, Principal Investigator, Head Endoscopy Unit, Valduce Hospital, Valduce Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 29052018_LCI
Record Dates: First submitted 2018-09-18; First posted 2018-10-01 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Colon Adenoma; Colonic Polyp
Keywords: adenoma detection rate; Linked Color Imaging; colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCI (Experimental): Linked Color Imaging
  Interventions: Device: Linked Color Imaging
- WL (Active Comparator): White Light
  Interventions: Device: Linked Color Imaging

INTERVENTIONS:
Device: Linked Color Imaging — Use of narrow band imaging with LCI for colon inspection during both insertion and withdrawal phase of colonoscopy

SUMMARY:
Linked color imaging (LCI) is newly developed image-enhancing endoscopy technology that differentiates the red color spectrum more effectively than white light imaging thanks to its optimal pre-process composition of light spectrum and advanced signal processing. This technology, combined in the latest generation Fujifilm's endoscopes (Fujifilm Co, Tokyo, Japan) with new high-performance LED illumination system, enhances the visibility of colonic mucosal vessels and might increase the detection rate of colorectal polyps. Data available regarding colorectal polyp or adenoma detection with LCI are encouraging but are scanty and limited to back-to back studies.

This two parallel arms, randomized, multicenter trial is aimed at evaluating whether LCI is superior to WL endoscopy in terms of adenoma detection

DETAILED DESCRIPTION:
50-75 years-old subjects participating in the regional screening program undergoing their first colonoscopy following a positive immunochemical fecal occult blood test (FIT) and meeting all eligibility criteria are randomised 1:1 to LCI (LCI group) or WLI (WL) during insertion and withdrawal phase of colonoscopy. A randomisation list for each participating center was produced by the coordinating center via computer-generated treatment code list. Randomisation is stratified by gender, age (50-60, 61-729 years) and screening history (first vs subsequent test) through an online centralised study database.All procedures are performed with a high-definition ELUXEO 700 series videocolonscopes with or without magnification (EC-760R, EC-760ZP, FUJIFILM Co., Tokyo).

The primary outcome measure is the ADR, defined as the proportion of participants with at least one adenoma (per-patient analysis).

ELIGIBILITY:
Inclusion Criteria:

* 50-75 years-old subjects participating in the regional screening program undergoing their first colonoscopy following a positive immunochemical fecal occult blood test (FIT)

Exclusion Criteria:

* subjects not eligible for invitation in the screening program (colonoscopy already performed in the previous 5 years, personal history of CRC, colonic adenomas or IBD, severe comorbidity, including end-stage cardiovascular, pulmonary, liver or renal disease)
* patients with inadequate bowel preparation (defined as Boston Bowel Preparation Scale > 2 in any colonic segment)
* patients with previous colonic resection
* patients on antithrombotic therapy, precluding polyp resection
* patients who were not able or refused to give informed written consent.

Ages: 50 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Adenoma Detection Rate | 1 year
  proportion of participants with at least one adenoma (per-patient analysis)

SECONDARY OUTCOMES:
advanced adenoma detection rate | 1 year
  proportion of participants with at least one advanced adenoma
mean number per subject of polyps, adenomas, advanced adenomas and sessile serrated lesions | 1 year
  total number of detected lesions in each group divided by the total number of participants
Withdrawal time | 1 year
  time for mucosal inspection only

CONTACTS AND LOCATIONS:
Overall Officials: Franco Radaelli, MD, Principal Investigator — Valduce Hospital, Como
Locations (1):
- Gastroenterology Unit, Valduce Hospital, Como, Italy

REFERENCES:
- [Derived] Paggi S, Radaelli F, Senore C, Maselli R, Amato A, Andrisani G, Di Matteo F, Cecinato P, Grillo S, Sereni G, Sassatelli R, Manfredi G, Alicante S, Buscarini E, Canova D, Milan L, Pallini P, Iwatate M, Rondonotti E, Repici A, Hassan C. Linked-color imaging versus white-light colonoscopy in an organized colorectal cancer screening program. Gastrointest Endosc. 2020 Sep;92(3):723-730. doi: 10.1016/j.gie.2020.05.044. Epub 2020 Jun 2. PMID 32502550